CLINICAL TRIAL: NCT03180710
Title: A Double-blinded, Randomised, Four-period Crossover Euglycemic Clamp Trial Investigating the Dose-linearity of BioChaperone® Combo 75/25 and the Safety at Three Different Doses in Subjects With Type 2 Diabetes
Brief Title: A Trial to Investigate the Dose-linearity of BioChaperone® Combo 75/25 and the Safety at Three Different Doses in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT025
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BioChaperone® Combo 75/25 at 0.6 U/kg (Experimental): Single subcutaneous injection of 0.6 U/kg
  Interventions: Drug: BioChaperone® Combo 75/25 at 0.6 U/kg
- BioChaperone® Combo 75/25 at 0.8 U/kg (Experimental): Single subcutaneous dose of 0.8 U/kg
  Interventions: Drug: BioChaperone® Combo 75/25 at 0.8 U/kg
- BioChaperone® Combo 75/25 at 1.0 U/kg (Experimental): Single subcutaneous dose of 1.0 U/kg
  Interventions: Drug: BioChaperone® Combo 75/25 at 1.0 U/kg
- Humalog® Mix25 at 0.8 U/kg (Active Comparator): Single subcutaneous dose of 0.8 U/kg
  Interventions: Drug: Humalog® Mix25 at 0.8 U/kg

INTERVENTIONS:
Drug: BioChaperone® Combo 75/25 at 0.6 U/kg — Injection of BioChaperone® Combo 75/25 at 0.6 U/kg
  Arms: BioChaperone® Combo 75/25 at 0.6 U/kg
Drug: BioChaperone® Combo 75/25 at 0.8 U/kg — Injection of BioChaperone® Combo 75/25 at 0.8 U/kg
  Arms: BioChaperone® Combo 75/25 at 0.8 U/kg
Drug: BioChaperone® Combo 75/25 at 1.0 U/kg — Injection of BioChaperone® Combo 75/25 at 1.0 U/kg
  Arms: BioChaperone® Combo 75/25 at 1.0 U/kg
Drug: Humalog® Mix25 at 0.8 U/kg — Injection of Humalog® Mix25 at 0.8 U/kg
  Arms: Humalog® Mix25 at 0.8 U/kg

SUMMARY:
This is a bicentric, double-blinded, randomised, four-period crossover phase 1 trial, using automated 30-hour euglycemic clamp in subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a bicentric, double-blinded, randomised, four-period crossover phase 1 trial, using automated 30-hour euglycemic clamp in subjects with type 2 diabetes mellitus.

Each subject will be randomly allocated to a sequence of four treatments, three single doses of BioChaperone® Combo 75/25 (0.6 U/kg, 0.8 U/kg or 1.0 U/kg) and one single dose of Humalog® Mix25 at 0.8 U/kg on four separate dosing visits.

Subjects will come in a fasted state to the clinical trial centre in the morning of each dosing day and stay at the clinical trial centre until the 30-hour clamp procedures have been terminated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18-70 years (both inclusive)
* Type 2 diabetes mellitus (as diagnosed clinically) for ≥ 12 months
* HbA1c level between 6.5% and 9.0 % (both inclusive)
* Body mass index between 20.0 and 40.0 kg/m2 (both inclusive)
* Body weight <= 125.0 kg at the screening visit
* Insulin-treated subjects. Total insulin dose of <= 1.2 (I)U/kg/day

Exclusion Criteria:

* Type 1 diabetes mellitus
* Known or suspected hypersensitivity to IMP(s) or related products
* Previous participation in this trial. Participation is defined as randomised.
* Receipt of any medicinal product in clinical development within 60 days before randomisation in this trial.
* Clinically significant abnormal values for haematology, biochemistry, coagulation, or urinalysis as judged by the Investigator considering the underlying disease.
* Supine blood pressure at screening (after resting for at least 5 min in supine position) outside the range of 90-160 mmHg systolically or 50-95 mmHg diastolically (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial); symptoms of arterial hypotension and/or a heart rate at rest outside the range of 50-90 beats per minute. This exclusion criterion also pertains to subjects being on anti-hypertensives.
* Women of child bearing potential not willing to use contraceptive methods.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
AUC last_total | From 0 to 30 hours
  Area under the plasma insulin concentration-time curve from t=0 to the last measured total insulin plasma concentration above LLOQ. The total insulin concentration is the sum of lispro and basal concentrations.
Cmax_total | From 0 to 30 hours
  Maximum observed plasma insulin total concentration

SECONDARY OUTCOMES:
AUCGIR 0-last (mg/kg) | From 0 to 30 hours
  Area under the glucose infusion rate curve from 0 hours until the end of clamp
GIRmax (mg/kg/min) | From 0 to 30 hours
  Maximum glucose infusion rate
tGIRmax | From 0 to 30 hours
  Time to maximum glucose infusion rate
Adverse Events | Up to 102 days (maximum duration of subject's participation)
Local tolerability: number of injection site reaction | Up to 102 days (maximum duration of subject's participation)
  Frequency of injection site reaction in each arm.
Number of hypoglycaemic events in each treatment arm | Up to 102 days (maximum duration of subject's participation)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: No